CLINICAL TRIAL: NCT07078942
Title: Effect of Preoperative Prophylactic Intravenous Tranexamic Acid on Perioperative Blood Loss in Pregnant Women Undergoing Cesarean Section : A Randomized Controlled Trial
Brief Title: Prophylactic Intravenous Tranexamic Acid on Perioperative Blood Loss in Pregnant Women Undergoing Cesarean Section
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Vorapong Phupong, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0127/68; COA 0685/2025 (Other: Chulalongkorn University)
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Pregnant Women Undergoing Cesarean Delivery
Keywords: tranexamic acid; blood loss; pregnant women; cesarean delivery
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Active Comparator): Tranexamic acid (1 g) 20 ml intravenous preoperation
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Normal saline 20 ml intravenous preoperation
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic Acid 1 g intravenous preoperation
  Arms: Tranexamic acid
Other: Placebo — normal saline 20 ml intravenous preoperation
  Arms: Placebo

SUMMARY:
The purpose of this study is to asses the effect of preoperative prophylactic intravenous tranexamic acid on perioperative blood loss in pregnant women undergoing cesarean section

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with gestational age 37-42 weeks
* undergoing cesarean delivery with indication as follows: placenta previa, severe preeclampsia, myoma uteri, fetal macrosomia, polyhydramnios, grand multiparity ≥ 5 deliveries, prolonged labor, etc.

Exclusion Criteria:

* history of allergy to tranexamic acid
* history of venous thromboembolism (Deep vein thrombosis, Pulmonary embolism)
* history of arterial thrombosis (Myocardial infarction, Stroke)
* history of seizure, convulsion
* have underlying of cardiovascular, renal or liver disease
* using of antiplatelet or anticoagulant within 1 week before operation
* placenta accreta spectrum
* abruptio placenta
* Eclampsia or HELLP (Hemolysis Elevated Liver Low Platelet) syndrome
* Failed operative vaginal delivery
* Multifetal gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 98 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood loss | From enrollment to the end of operation
  blood loss in ml

SECONDARY OUTCOMES:
early postpartum hemorrhage | From starting operation to 24-hour postoperation
  percentage of early postpartum hemorrhage
delayed postpartum hemorrhage | From starting operation to 6 weeks postpartum
  percentage of delayed postpartum hemorrhage
Adverse effects | from enrollment to 6 weeks postpartum
  percentage of adverse effects
Neonatal outcomes | from starting operation to 10 minutes after birth
  Apgar scores (0 is the minimum value and 10 is maximum value, and higher scores mean a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Vorapong Phupong, M.D., Study Director — Chulalongkorn University
Locations (1):
- Department of Obstetrics and Gynecology, Faculty of Medicine, Chulalongkorn University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Waiting for the permission from IRB

REFERENCES:
- [Background] Sentilhes L, Senat MV, Le Lous M, Winer N, Rozenberg P, Kayem G, Verspyck E, Fuchs F, Azria E, Gallot D, Korb D, Desbriere R, Le Ray C, Chauleur C, de Marcillac F, Perrotin F, Parant O, Salomon LJ, Gauchotte E, Bretelle F, Sananes N, Bohec C, Mottet N, Legendre G, Letouzey V, Haddad B, Vardon D, Madar H, Mattuizzi A, Daniel V, Regueme S, Roussillon C, Benard A, Georget A, Darsonval A, Deneux-Tharaux C; Groupe de Recherche en Obstetrique et Gynecologie. Tranexamic Acid for the Prevention of Blood Loss after Cesarean Delivery. N Engl J Med. 2021 Apr 29;384(17):1623-1634. doi: 10.1056/NEJMoa2028788. PMID 33913639
- [Background] Pacheco LD, Clifton RG, Saade GR, Weiner SJ, Parry S, Thorp JM Jr, Longo M, Salazar A, Dalton W, Tita ATN, Gyamfi-Bannerman C, Chauhan SP, Metz TD, Rood K, Rouse DJ, Bailit JL, Grobman WA, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Tranexamic Acid to Prevent Obstetrical Hemorrhage after Cesarean Delivery. N Engl J Med. 2023 Apr 13;388(15):1365-1375. doi: 10.1056/NEJMoa2207419. PMID 37043652
- [Background] Cheema HA, Ahmad AB, Ehsan M, Shahid A, Ayyan M, Azeem S, Hussain A, Shahid A, Nashwan AJ, Mikus M, Lagana AS. Tranexamic acid for the prevention of blood loss after cesarean section: an updated systematic review and meta-analysis of randomized controlled trials. Am J Obstet Gynecol MFM. 2023 Aug;5(8):101049. doi: 10.1016/j.ajogmf.2023.101049. Epub 2023 Jun 11. PMID 37311484
- [Background] Angolile CM, Max BL, Mushemba J, Mashauri HL. Global increased cesarean section rates and public health implications: A call to action. Health Sci Rep. 2023 May 18;6(5):e1274. doi: 10.1002/hsr2.1274. eCollection 2023 May. PMID 37216058
- See also: Related Info — https://www.who.int/publications/i/item/WHO-RHR-17.21
- See also: Related Info — https://www.acog.org/news/newsreleases/2017/09/acog-expands-recommendations-to-treat-postpartum-hemorrhage.